CLINICAL TRIAL: NCT02063009
Title: Measurement of Cardiac Index by Transpulmonary Thermodilution Using an Implanted Central Venous Access Port: a Prospective Study in Patients Scheduled for Oncologic High-risk Surgery
Brief Title: Measurement of Cardiac Index Using an Implanted Central Venous Access Port in Patients Scheduled for Oncologic High-risk Surgery
Acronym: ThermoD-PAC
Status: Completed | Type: Observational
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A00003-40; 2012/1836 (Other: CSET number)
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Oncologic High-risk Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients scheduled for oncologic high-risk surgery

SUMMARY:
Perioperative hemodynamic optimization requires monitoring adapted to the risks of the surgery and the patient. We currently use a local hemodynamic protocol based on the data of the literature. According to this protocol, specific patients may require cardiac index and central venous oxygen saturation monitoring. We chose to monitor the cardiac index (CI) with the transpulmonary thermodilution technique (TPTD) (PiCCO, Pulsion Medical System, Munich, Germany). The technique is based on the injection of a cooled bolus of saline into a central vein with a central venous catheter (CVC). The variation of temperature is measured with an arterial femoral catheter and allows the assessment of the cardiac output according to Stewart-Hamilton's theory. Many studies showed the reliability of this technique.

In our institute, most of the patients are fitted with a port for chemotherapy or parenteral nutrition. When PiCCO monitoring is necessary, a central venous catheter is inserted on the opposite side of the permanent implantable venous port. Indeed, insertion of the CVC can be more difficult because of the port. It may be interesting to use the port for TPTD in order to avoid the insertion of a new CVC. This would be possible only if the measurement of CI by the port was as reliable as the classical measurement with a CVC.

DETAILED DESCRIPTION:
The aim of this study was to assess whether measurement of the CI by TPTD was possible and reliable via the port. We conducted a prospective study comparing the measurement of the CI by TPTD before and after fluid challenge via the port versus the CVC.

ELIGIBILITY:
Inclusion Criteria:

* presence of port
* scheduled surgery with perioperative optimization requirement according to the local hemodynamic protocol
* oral consent of the patient after oral and written information

Exclusion Criteria:

* age inferior to 18
* Contraindication or failure to the insertion of the CVC
* Contraindication to the use of the port : local or general infection suspected or proved, absence of blood backflow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for oncologic high-risk surgery
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Estimation of the reliability of the measurement of the variations of the CI during fluid challenge | measurement of the CI hourly, up to 3 hours by TPTD before and after fluid challenge via the port versus the CVC.
  Measurements will be realized as described:
  * hourly: TPTD will be realized to calibrate the measurement of CI
  * Before and after fluid challenge (250 ml of colloid when hemodynamic indicators will be in favour of hypovolemia (pulse pressure variation (PPV) > 15% and variation of CI > 10%)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Eghiaian, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Suria S, Wyniecki A, Eghiaian A, Monnet X, Weil G. Measurement of cardiac index by transpulmonary thermodilution using an implanted central venous access port: a prospective study in patients scheduled for oncologic high-risk surgery. PLoS One. 2014 Aug 19;9(8):e104369. doi: 10.1371/journal.pone.0104369. eCollection 2014. PMID 25136951